CLINICAL TRIAL: NCT03791151
Title: Effect of Copper Transporter-1 Genetic Polymorphism on Platinum Based Chemotherapy Response in Advanced Non-Small Cell Lung Cancer Patients
Brief Title: Pharmacogenetics in Non Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yara Sayed Abdulwahid, Clinical Pharmacist, Ain Shams University
Other Study IDs: ASU309
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Pharmacogenetics; Lung cancer; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the effect of genetic polymorphism in the membrane copper transporter 1 protein [CTR1; encoded by the solute carrier family 31 member 1 gene (SLC31A1 gene)] and its genetic expression levels on the clinical outcome of cisplatin-based regimen used in the treatment of Non-Small Cell Lung Cancer (NSCLC) in terms of :

* Treatment response : partial response (PR) / complete response (CR) and Progression-free survival (PFS)
* Treatment resistance : stationary disease (SD) or progressed disease
* Frequency and severity of regimen related toxicity

DETAILED DESCRIPTION:
The cisplatin-based regimen is an effective treatment for advanced NSCLC, showing significant beneficial outcomes such as prolong survival, improve clinical symptoms, and improve quality of life (QOL) . Although platinum-based therapy shows several benefits, but the five-year survival rate still less than 20%.

Pt resistance is an inevitable occurrence with rare exception. Aside from germ cell tumors, metastatic solid tumors are generally thought to be incurable with cytotoxic chemotherapy due to the development of resistance and subsequent disease progression.

Despite the multifactorial nature of Cisplatin resistance, intracellular accumulation of Pt appears to be a major source of drug resistance . Reduced intracellular drug accumulation is one of the most consistently identified features of cisplatin-resistant cells.

Many evidences indicated that alteration of copper transporter protein 1 (CTR1) which is the major plasma membrane transporter responsible for platinum uptake, was associated with platinum sensitivity and toxicity.

Genetic polymorphisms of CTR1 also have effects to platinum treatment response. Therefore, CTR1 might be a potential prognostic factor for survival in cancer patients underwent chemotherapy and a treatment target for overcoming platinum resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with immunohistochemically and pathologically confirmed non- small cell lung cancer (NSCLC).
2. ECOG PS 0-2.
3. Chemotherapy naïve.
4. Age >18 years.
5. Adequate bone marrow reserve.

Exclusion Criteria:

1. Presence of central nervous system metastases.
2. Inadequate liver function (bilirubin > 1.5 times upper normal limit [ULN] and alanine transaminase [ALT] or aspartate transaminase [AST] > 3.0 ULN or up to 5.0 UNL in the presence of hepatic metastases).
3. Inadequate renal function (creatinine > 1.25 times ULN, creatinine clearance < 50mL/min).
4. Serious comorbid systemic disorder incompatible with the study.
5. Second primary malignancy (except in situ carcinoma of the cervix, adequately treated basal cell carcinoma of the skin, T1 vocal cord cancer in remission, or prior malignancy treated more than 5 years prior to enrollment without recurrence).
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed with immunohistochemically and pathologically confirmed non- small cell lung cancer (NSCLC).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Tumor response and resistance | 1 year
  will be evaluated after the third (initial evaluation response) and the sixth (confirmation of initial response) chemotherapy cycle according to the new Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1.5 years
  defined as the time from day 1 of chemotherapy to the day of documented disease progression or death.
Regimen related toxicity | 1.5 years
  1. Hematologic toxicity (anemia, neutropenia, and thrombocytopenia) 2. Nephrotoxicity 3. Ototoxicity 4. Neurotoxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University's Hospital, Cairo, Egypt

REFERENCES:
- [Background] Blair BG, Larson CA, Safaei R, Howell SB. Copper transporter 2 regulates the cellular accumulation and cytotoxicity of Cisplatin and Carboplatin. Clin Cancer Res. 2009 Jul 1;15(13):4312-21. doi: 10.1158/1078-0432.CCR-09-0311. Epub 2009 Jun 9. PMID 19509135
- [Background] Roco A, Cayun J, Contreras S, Stojanova J, Quinones L. Can pharmacogenetics explain efficacy and safety of cisplatin pharmacotherapy? Front Genet. 2014 Nov 14;5:391. doi: 10.3389/fgene.2014.00391. eCollection 2014. PMID 25452763
- [Background] Xu X, Ren H, Zhou B, Zhao Y, Yuan R, Ma R, Zhou H, Liu Z. Prediction of copper transport protein 1 (CTR1) genotype on severe cisplatin induced toxicity in non-small cell lung cancer (NSCLC) patients. Lung Cancer. 2012 Aug;77(2):438-42. doi: 10.1016/j.lungcan.2012.03.023. Epub 2012 Apr 17. PMID 22516052
- See also: The role of the mammalian copper transporter 1 in the cellular accumulation of platinum-based drugs. — https://www.ncbi.nlm.nih.gov/pubmed/18996970